CLINICAL TRIAL: NCT00862368
Title: Sustaining Cessation in Smokers With Kids With Asthma
Brief Title: Sustaining Smoking Cessation in Smokers With Kids With Asthma
Acronym: PAQS2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other); University of California, Berkeley (Other); RTI International (Other); Rhode Island Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Belinda Borrelli, Professor of Psychiatry and Human Behavior, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01HL062165-09 (NIH); R01HL062165 (NIH)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Asthma; Smoking Cessation
Keywords: Motivational Interviewing; Pediatric Asthma; Smoking Cessation; Environmental Tobacco Smoke; Second hand smoke; Biomarker; Asthma; Asthma Education; Family Intervention; Smoking; Nicotine Patch; Parents; Caregivers; Child Wellness
MeSH Terms: conditions — Asthma; Smoking Cessation; Smoking | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PAM -Enhanced/Asthma (Experimental): The PAM-Enhanced/Asthma group: 2 in-home visits that included asthma education consistent with NIH recommendations (NIH, NAEPP, 1997) and smoking cessation counseling. Consistent with Motivational Interviewing (MI), smoking was broached in a non-judgmental manner and as another trigger for asthma. Feedback was given on expired air Carbon Monoxide (CO) levels of the smoker (to increase personal perception of risk) and the amount of smoke exposure to the child (to increase risk perception to the child). 6 phone calls were then provided over the next 4 months that focused on asthma education, a second round of feedback on the child's ETS exposure, and smoking cessation counseling. MI was used at all contacts. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Interventions: Behavioral: PAM; Behavioral: PAM-Enhanced/Asthma Counseling Phone Calls
- PAM-Asthma (Active Comparator): The PAM-Asthma arm received the same in-home counseling visits as PAM-Enhanced/Asthma. The 6 counseling phone calls were different from those received by PAM-Enhanced/Asthma, and included only an asthma follow-up and discussion of a child wellness topic. Smoking cessation was not discussed and additional feedback on ETS samplers was not provided. Motivational Interviewing approaches were used in all in-home and phone counseling. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Interventions: Behavioral: PAM
- PAM-Healthy (Active Comparator): The PAM-Healthy arm received the same in-home counseling visits as PAM and PAM Enhanced but asthma information was replaced with child wellness topics. The 6 counseling phone calls were the same timing and duration as the other two groups (six, 15 minutes calls, over four months) focused on a child wellness topic. Smoking cessation or sampler feedback was not discussed. Motivational Interviewing approaches were used in all in-home and phone counseling. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Interventions: Behavioral: PAM; Behavioral: Follow-Up Phone Calls - Child Wellness Topic

INTERVENTIONS:
Behavioral: PAM — Visit 1 included asthma education (or child wellness for healthy children), expired air carbon monoxide feedback, Motivational Interviewing, and techniques to accelerate the participants readiness to quit. Visit 2 included a follow up on the child's asthma (PAM and PAM-Enhanced only), assessing the smoker's motivation to quit, feedback on CO readings and air sampler results (smoke exposure to the child), risks of smoking, and benefits of quitting. Counselors employed Motivational Interviewing techniques. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Other Names: PAM-Asthma; PAM-Enhanced/Asthma; PAM-Healthy; PAQS; Asthma Education; Smoking Cessation Counseling; Motivational Interviewing
Behavioral: PAM-Enhanced/Asthma Counseling Phone Calls — PAM-Enhanced/Asthma counseling calls were made over the 4 months following in-home counseling and focused on: 1) checking in on the child's asthma, 2) motivating quit attempts, and 3) preventing relapse among quitters. The final phone call (#6) included feedback on the 2nd set of air samplers placed in the home and with the child after phone call 5. Only the PAM-Enhanced/Asthma condition received this 2nd round of ETS feedback. A printed feedback report was provided to participants. If still smoking, counseling focused on ETS reduction and motivation to change. If quit, counseling focused on reinforcement of successful behavior change and motivation to stay quit. Motivational Interviewing techniques were used. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Other Names: Smoking Cessation Counseling; Phone Counseling; Motivational Interviewing
  Arms: PAM -Enhanced/Asthma
Behavioral: Follow-Up Phone Calls - Child Wellness Topic — Over the 4 months following in-home counseling visits, subjects in the PAM-Asthma and PAM-Healthy conditions received 6 phone calls that included an asthma check-in (PAM-Asthma only) and discussion of a child wellness topic. Counselors employed Motivational Interviewing techniques. Free nicotine patch tx was given if they were ready to quit within 30 days.
  Other Names: PAM-Asthma; PAM-Healthy; Child Wellness; Phone Counseling; Motivational Interviewing
  Arms: PAM-Healthy

SUMMARY:
Parents of Asthmatics Quit Smoking (PAQS-2) is a randomized controlled trial of a smoking cessation intervention for parents who smoke. Children had either a diagnosis of asthma (and an asthma emergency within the past 3 months) or were healthy (and had no medical conditions in the past 3 months). The study intervention aimed to help parents (or caregivers) quit smoking and reduce children's second hand smoke exposure. Participants received 2 home counseling sessions with asthma education (if they had a child with asthma), child wellness (if they had a healthy child) and smoking cessation counseling (including objective feedback on how much smoke the child was exposed to). Parents of children with asthma were then randomized into 2 groups; one group received 6 counseling phone calls focused on motivating smoking cessation and a second round of feedback on smoke exposure (Enhanced). The other groups received six calls focused on asthma (PAM asthma group) or child wellness (Healthy group). We had 2 primary aims. First, to explore the "teachable moment" we compared quit rates between the parents of children with asthma to the parents of healthy children. We hypothesized that the Asthma group would have significantly greater quit rates than the Healthy group and lower levels of environmental tobacco smoke in the home. We also hypothesized that parents who smoke and have children with asthma would have greater changes in the variables associated with teachable moment compared to parents who smoke and have a healthy child. --- The second primary aim focused on the parents of children with asthma. We assessed the effectiveness of adding telephone smoking cessation counseling to the 2 home counseling visits. For this, we compared the 2 groups of randomized subjects: those who received 6 counseling calls and feedback on smoke exposure (PAM-Enhanced) and those who received 6 counseling calls focused on asthma education (PAM-Asthma). We hypothesized that the PAM-Enhanced group would have significantly greater quit rates than the PAM-Asthma group, lower likelihood of smoking relapse, and lower levels of environmental tobacco smoke in the home. We also explored the hypothesized role of precaution effectiveness (i.e. quitting smoking will be associated with benefits for self and child) and self-efficacy for quitting as mediators of the effectiveness of PAM-Enhanced/Asthma. A third aim was to compare asthma symptoms over time between the two groups.

DETAILED DESCRIPTION:
Asthma is one of the most common pediatric diseases affecting 6.7 million children and adolescents (Akinbami et al 2009). Asthma is a leading cause of hospitalizations, emergency department visits, school absences, and activity restriction for youth (ALA, 2011; Taylor et al., 1992; Weiss et al., 1992). Smoking is the leading cause of preventable morbidity and mortality as 443,000 deaths are attributable to smoking each year (CDC, 2012).

This study had two aims that built on the results of a previous study (Borrelli et al., 2002): 1) to characterize the cognitive, affective, and behavioral changes associated with the Teachable Moment (TM), and 2) to test whether or not an extended intervention augments quit rates and prevents relapse over and above a previous theory-based smoking cessation intervention for low-income caregivers of children with asthma (Borrelli et al., 2002).

In our study, we viewed the provision of objectivefeedback about the child's exposure to ETS as necessary to link the caregiver's smoking with the child's asthma. It was hypothesized that providing feedback within the context of heightened awareness of the child's health constitutes the teachable moment. The first aim of this study was to examine, in two populations, the effect of an intervention based on The Precaution Adoption Model (PAM) (Weinstein, 1988), in which Motivational Interviewing and biomarker feedback (smoker's CO level and child's ETS exposure) were used to increase risk perception to self and child. Our populations were: 1) smokers whose child with asthma had an acute exacerbation (PAM-Asthma) and 2) smokers who had a healthy child (PAM-Healthy).

The second aim was to test the effect of increasing the intensity of our original theory-based intervention, PAM, by adding telephone counseling that focuses on motivating and sustaining quit attempts. Though our previous study demonstrated excellent quit rates in the short term (at 2 month follow-up), there was a dramatic decrease in abstinence by 6 months. Therefore, caregivers of kids with asthma were randomized to either 1) PAM-Asthma: our original intervention plus six contact control calls focusing on the child's asthma and child wellness (diet, exercise, safety, etc.) or 2) PAM-Enhanced/Asthma: our original intervention plus six counseling calls that focus on the child's asthma, motivating quit attempts, and preventing relapse. Precaution effectiveness (belief that quitting will improve one's own and the child's health) and self-efficacy were the primary intervention targets during the PAM-Enhanced/Asthma calls.

A. Primary Aims

Aim 1: To assess the cognitive, affective, and behavioral changes involved in the "teachable moment" by examining those who receive PAM and have children with asthma (PAM-Asthma) vs. those who receive PAM and have healthy children (PAM-Healthy).

Hypothesis 1.1: PAM-Asthma will, at follow-ups, have significantly greater quit rates than PAM-Healthy (7-day point prevalence abstinence, 30 day abstinence) and lower levels of ETS in the home.

Hypothesis 1.2: Parents who smoke and have children with asthma (PAM-Asthma) will have greater changes in the variables hypothesized to be associated with teachable moment (perceived risk, affect, self-concept) vs. parents who smoke and have a healthy child (PAM-Healthy). We are also exploring the mediational role of these factors on outcome.

Aim 2: Among the parents of children with asthma, to assess the effectiveness adding telephone counseling to our previously tested intervention, PAM, (PAM-Enhanced/Asthma) vs. PAM plus contact control (PAM-Asthma).

Hypothesis 2.1. PAM-Enhanced/Asthma will, at follow-ups, have significantly greater quit rates than PAM-Asthma (7 day point prevalence abstinence, 30 day abstinence), lower likelihood of relapse, and lower levels of ETS in the home.

Hypothesis 2.2. Explore the hypothesized role of precaution effectiveness (i.e., quitting smoking will be associated with benefits for self and child) and self-efficacy for quitting as mediators of the effectiveness of (PAM-Enhanced/Asthma). We also plan to explore the effect of important moderating variables (demographics, social support, depressed mood) on smoking outcomes.

B. Secondary Aims:

Aim 3: To assess differences between PAM-Enhanced/Asthma and PAM-Asthma groups in asthma morbidity and health care utilization among children with asthma.

Hypothesis 3.1: PAM-Enhanced/Asthma will have lower levels of functional morbidity due to asthma (i.e., fewer symptoms and less activity limitations) vs. PAM-Asthma.

Hypothesis 3.2: PAM-Enhanced/Asthma will have lower levels of health care utilization including fewer hospital days for asthma, fewer urgent care visits for asthma, and fewer prescription refills for quick-relief asthma medications vs. PAM-Asthma.

C. Study Design

This was a three group design with 2 group comparisons. In order to test Aim 1 (Teachable Moment) smokers with kids with asthma (PAM-Asthma) were compared to smokers with healthy kids (PAM-Healthy) on their cognitive, affective, and behavioral changes before and immediately after receiving feedback on the child's smoke exposure. Both groups received home-based smoking cessation counseling (PAM), and six contact control calls focused on child wellness or asthma education. In order to test Aim 2, improving and sustaining the smoking cessation rates, smokers with kids with asthma were randomly assigned to receive to either PAM + six contact control calls (PAM-Asthma) or PAM + six counseling calls that focused on building precaution effectiveness and self-efficacy (PAM-Enhanced).

ELIGIBILITY:
Inclusion Criteria: In order to be included in the study, participants had to:

* be caregivers for a child (defined as having the child in the home for at least 4 hours per week) between the ages of 3 and 17,
* be current, regular smokers (at least 3 cigarettes per day for the past year)
* be over age 18
* speak and understand English
* have a telephone
* agree to participate in all phases of the study
* have a child with a diagnosis of asthma (asthma groups only)

Exclusion Criteria:

* if the index child had asthma, child DID NOT have a urgent care/emergency room/hospital visit within 90 days of the first intervention visit
* if the index child was healthy, child DID have a urgent care/emergency room/hospital visit within 90 days of the first intervention visit and had no diagnosis of asthma (or other children in the home with asthma)
* had children with other significant pulmonary disease
* the index child spent less than 4 hours in the home per week
* caregiver exclusively used another form of tobacco (not cigarettes)
* using any form of Nicotine replacement therapy
* using medications to quit smoking
* in a quit smoking program
* another member of family is participating in program
* currently pregnant or planning to become pregnant

While we did offer the intervention to all smokers in the home, only the caregiver that spent the most time with the child was included in the formal study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 573 (Actual)
Dates: Start 2005-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Smoking Status | 2 months after the end of home visits; after the end of the phone calls (4 months). The 6 month follow-up occurred approximately 2 months after the four month assessment and the 12 month assessment occurred 6 months after the 6 month assessment.
  Smoking Status was assessed at all follow-up assessments. Seven-day point prevalence abstinence (no smoking at all in the previous seven days, not even a puff) and 30 day point-prevalence abstinence (no smoking at all in the previous 30 days, not even a puff) were used as dependent variables. CO Verification: Those participants who reported a smoking status of "Quit" at follow-up assessments were tested for carbon monoxide levels using a exhaled breath analyzer. Those with Carbon Monoxide readings <=10 ppm were considered abstinent.

SECONDARY OUTCOMES:
Environmental Tobacco Smoke, Self-Report | Baseline, and 2 mos after the end of home visits; after the end of phone calls (4 mos). The 6 month follow-up was approximately 2 months after the 4 month assessment and the 12 month assessment occurred 6 mos after the 6 month assessment.
  A self-report questionnaire (Matt, Hovell et al., 2000) was administered using a structured interview designed to elicit reliable memory-based reports of the participant's own smoking rate as well as their report of others' smoking rates while in the home. The interview contains questions that assess the total, average, least, and greatest number of cigarettes smoked in the home, in the car and away from home. Another questionnaire, The Environmental Tobacco Smoke Survey, assessed whether or not participants' had smoking bans in their home and car, and their readiness to implement these bans.
Environmental Tobacco Smoke: Air Samplers | Placed at baseline and collected after 7 days of exposure; Placed after phone call 5 (approximately 3.5 months after Intervention Visit 2) and collected after 7 days exposure.
  ETS was objectively measured with passive nicotine air samplers that utilize nicotine as a tracer for ETS. Samplers use a filter treated with sodium bisulfate (weak acid) which reacts with nicotine(a weak base) to form a stable salt. The filter is contained in a 4 cm polystyrene cassette, which has a membrane filter as a windscreen. For each participant, one sampler was placed in the room in which the child spends the most time and one was worn by the child (at baseline and at after the 5th follow-up phone call for 7 days each). Samplers were analyzed by Co-I Hammond.
Asthma Morbidity | Baseline and 2 mos after the end of home visits; after the end of phone calls (4 mos). The 6 month follow-up was approximately 2 months after the 4 month assessment and the 12 month assessment occurred 6 mos after the 6 month assessment.
  Functional morbidity due to asthma was measured using the Asthma Assessment Form, adapted from the Functional Severity scale by Rosier et al. (1994). Questions assess the child's asthma symptoms over the past month, and assess how asthma has impacted limitations in general activity, school attendance, and sports participation for school-aged children. Questions about frequency of doctor visits, emergency room visits, hospitalizations, and medication use (including rescue inhaler, nebulizer, and steroid use) are also included.

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Borrelli, PhD, Principal Investigator — Brown University/The Miriam Hospital
Locations (5):
- United States (5):
  - St. Anne's Hospital, Fall River, Massachusetts
  - Memorial Hospital of RI, Pawtucket, Rhode Island
  - Hasbro Children's Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island

REFERENCES:
- [Background] Wagener TL, Gregor KL, Busch AM, McQuaid EL, Borrelli B. Risk perception in smokers with children with asthma. J Consult Clin Psychol. 2010 Dec;78(6):980-5. doi: 10.1037/a0021094. PMID 21114346
- [Derived] Borrelli B, McQuaid EL, Tooley EM, Busch AM, Hammond SK, Becker B, Dunsiger S. Motivating parents of kids with asthma to quit smoking: the effect of the teachable moment and increasing intervention intensity using a longitudinal randomized trial design. Addiction. 2016 Sep;111(9):1646-55. doi: 10.1111/add.13389. Epub 2016 May 17. PMID 27184343